CLINICAL TRIAL: NCT00091845
Title: An Exploratory Study of the Safety, Tolerability, Pharmacokinetics and Potential Effectiveness of AVI-4020 Injection in Patients Presenting With Presumptive Acute Neuroinvasive West Nile Virus (WNV) Disease
Brief Title: An Exploratory Study of AVI-4020 in Patients With Possible Acute Neuroinvasive West Nile Virus (WNV) Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to limited pool of eligble WNV patients
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVI-4020-14
Record Dates: First submitted 2004-09-17; First posted 2004-09-21 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: West Nile Fever
Keywords: West Nile Fever Myelitis; West Nile Fever Encephalitis; West Nile Fever Meningitis; West Nile Fever Meningoencephalitis
MeSH Terms: conditions — West Nile Fever

INTERVENTIONS:
Drug: AVI-4020 Injection

SUMMARY:
Although the serious form of West Nile Virus (WNV) disease, referred to as neuroinvasive disease, is rare, it can result in permanent disabilities and occasionally death. For patients who get this serious form of WNV disease, there are no approved specific treatment options.

The purpose of this study is to test a new drug, AVI-4020 Injection, in patients who are hospitalized with recent symptoms of this form of WNV disease. In this study, we will determine if the AVI-4020 treatment is safe. This will be accomplished by reviewing the results of laboratory tests and clinical signs and symptoms. Additionally, we will review the patient data for signs that AVI-4020 is providing any beneficial effects against WNV neuroinvasive disease.

DETAILED DESCRIPTION:
1. To evaluate the safety of intravenously administered (IV) AVI-4020 Injection every 12 hours for a total of ten doses over the course of study surveillance.
2. To evaluate the tolerability of intravenously administered AVI-4020 Injection every 12 hours for a total of ten doses over the course of study surveillance.
3. To evaluate the effectiveness of intravenously administered AVI-4020 Injection at 45 mg every 12 hours for ten doses, based on the neurological status of each study Subject as measured by a combination of the NIH stroke scale score and the Glasgow coma scale score.
4. To evaluate the robustness of the potential effectiveness of intravenously administered AVI-4020 Injection every 12 hours for ten doses over the course of 35 days of active surveillance, based on a variety of criteria, e.g., clinical, laboratory and/or neurophysiological results.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a positive serum or CSF ELISA MAC-IgM test indicating active/recent WNV infection, or the Subject resides in or has traveled to geographic areas with at least one of the following characteristics within the last seven days:

  1. Documented evidence of WNV infected mosquitoes or sentinel animals within the last 30 days
  2. Documented evidence of WNV infected dead animals within the last 30 days
  3. Documented human cases of WNV infection/disease within the last two weeks
* Subject is between >18 and <75 years of age.
* Subject has developed a febrile disease with new neurological findings <4 days prior to the current hospitalization.
* Subject has had an oral temperature of >38 degrees Celsius within 48 hours of study entry.
* Subject must have one or more of the following acute signs at the time of study entry:

  1. Signs of meningitis (nuchal rigidity)
  2. Signs of encephalitis (changes in mental status)
  3. Evidence of brainstem, cranial nerve, or cerebellar dysfunction
  4. Limb weakness.
* Subject must have a CSF examination within 48 hours of study entry showing:

  1. Absence of any organisms on Gram or fungal stains
  2. White blood cell count of > 4 per mm3 (corrected for significant red blood cell contamination)
  3. Ratio of CSF glucose: plasma glucose of >0.40; and CSF protein >30 mg/dL
* Subjects with reproductive potential must agree to practice adequate birth control methods to protect themselves and their partners from conception as defined below:

  1. Men with reproductive potential are eligible to participate if they use an acceptable method of contraception (such as a condom with spermicide).
  2. Women with childbearing potential are eligible to participate if they are surgically sterile (via hysterectomy or bilateral tubal ligation) at least one year post-menopausal, or are using an acceptable method of contraception (such as oral, topical, or injected contraception, IUD, Nuva-Ring®, or double barrier method such as diaphragm and condom with spermicide).

Exclusion Criteria:

* Subject (or family or legal guardian) requests Do Not Resuscitate or Do Not Intubate orders.
* Subject has multi-system organ failure at the time of screening or is not expected to survive the next 12 months due to another cause.
* Subject has a history of any vaccine administration <30 days prior to study entry.
* Subject has a possible history of traumatic neuritis <7 days prior to study entry (e.g., acupuncture, any needle-administered drugs, automobile accident, and/or blunt trauma).
* Subject is female and is pregnant or breastfeeding. (If the Subject is not postmenopausal or has not been surgically sterilized, a negative serum pregnancy test is required within 72 hours prior to the administration of the first dose of study drug.)
* Subject has any of the following clinically significant abnormal laboratory results:

  1. Serum creatinine greater than 3.0 mg/dL or study Subject requires hemodialysis
  2. Liver function tests twice the upper limit of normal
  3. Total bilirubin level twice the upper limit of normal
  4. PT or INR twice the upper limit of normal
* Documented presence of bacterial or non-WNV viral agents in CSF
* Principal Investigator is of the opinion that the Subject's medical condition(s) or state of mental health would prevent adherence to protocol requirements or hinder interpretation of clinical study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-11; Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessments will be based on evaluations of treatment emergent adverse events (TEAE), serious adverse events (SAE), serial clinical examinations, and serial conventional laboratory tests.

SECONDARY OUTCOMES:
A secondary endpoint is the potential effectiveness of AVI-4020 Injection based on the neurological status measured by a combination of the NIH Stroke Scale and the Glasgow Coma Score (GCS).